CLINICAL TRIAL: NCT05558397
Title: Effectiveness of Epidural Morphine and Ropivacaine Treatment for Abdominal Cancer Pain in Patients of Brazilian's Public Health System
Brief Title: Epidural Association of Morphine and Ropivacaine for Cancer Pain Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Alfenas (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Larissa Helena Lobo Torres Pacheco, PhD Professor, Universidade Federal de Alfenas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2.543.790
Record Dates: First submitted 2022-09-13; First posted 2022-09-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cancer Pain; Opioid Use; Cost Analysis; Palliative Care; Epidural Route; Morphine-ropivacaine Association; Quality of Life; Rational Use of Medication
MeSH Terms: conditions — Cancer Pain | interventions — Control Groups; Morphine

STUDY DESIGN:
Intervention Model Description: Control group: oral route morphine Intervention group: epidural route morphine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Oral Morphine) (Active Comparator): The control group will be composed of 15 patients who will receive oral drug treatment according to the Clinical Protocol and Therapeutic Guidelines for Chronic Pain of the Brazilian Ministry of Health. The drugs included in the treatment plan are morphine (60 mg/day), pregabalin (150 mg/day) and duloxetine (60 mg/day), available free of charge to the participating patients. The treatment will be carried out orally in a home environment.
  Interventions: Drug: Control Group (Oral morphine)
- Interventional Group (Epidural morphine) (Experimental): The intervention group will be composed of 15 patients who will undergo a surgical procedure for subcutaneous implantation of a catheter (Celsite ST304-19BBraun) that allows epidural administration of morphine and ropivacaine drugs. The treatment plan for such patients includes Patient Controlled Analgesia (PCA). Patients in this group will receive, via catheter, an anesthetic solution containing 2.0 mL of morphine (1.0 mg/mL), 3.0 mL of ropivacaine (7.5 mg/mL) and 5.0 mL of distilled water. For 24 hours after this application, if the patient continues to have pain, they may use a rescue dose of oral morphine of 10 mg.
  Interventions: Device: Interventional Group (Epidural morphine)

INTERVENTIONS:
Device: Interventional Group (Epidural morphine) — Implantation of an epidural catheter for administration of morphine and ropvacaine
  Arms: Interventional Group (Epidural morphine)
Drug: Control Group (Oral morphine) — Oral administration of morphine, pregabalin or duloxetin
  Arms: Control Group (Oral Morphine)

SUMMARY:
In 2012, more than 14 million cases of cancer were diagnosed worldwide, with the forecast for 2025 exceeding 20 million. Pain is the most critical symptom that accompanies cancer. The development of disease generates the need for oncological palliative care and adequacy of the structure by Public Health Care System. In this context, this study aims to evaluate an alternative to the treatment plans provided for in the Brazilian's Public Health Care System table. The objective is to carry out a cost-effectiveness analysis of the epidural administration of morphine and ropivacaine in patients with abdominal neoplasia, and pain that is difficult to clinically control, which leads to an improvement in the quality of life, functional conditions and survival of patients, and that reduces the cost to the Brazilian's Public Health Care System. This is a randomized clinical trial. Patients will be divided into two groups: control and intervention. The control group will receive oral treatment according to the Clinical Protocol and Therapeutic Guidelines for Chronic Pain of the Brazilian's Ministry of Health: morphine, pregabalin and duloxetine. The intervention group will receive an anesthetic solution containing morphine and ropivacaine for epidural administration through a surgically implanted catheter. Pain, quality of life, functional capacity and survival will be evaluated using the following instruments: Visual Analogue Scale; European Organization for Research and Treatment of Cancer Quality of Life Questionnaire "Core" 30; Karnofsky Performance Scale; Eastern Cooperative Oncology Group Scale; Palliative Performance Scale; and Palliative Prognosis Index. It is expected that, at the end of the study, the intervention group will represent a significant savings for the Public Health Care System, due to the decrease in the number of hospitalizations/day and the possible complications due to the lack of effectiveness of the oral treatment. It is expected that the results found will produce scientific support to disseminate the proposed treatment plan for Brazilian's Public Health Care System patients in palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years,
* both sexes
* diagnosed with abdominal neoplasia and with PPI < 2.0, which indicates a survival of at least 90 days
* have full cognitive conditions
* Patients must also have a caregiver with cognitive conditions.

Exclusion Criteria:

- Patients with technical incapacity to implant the catheter will be excluded, namely: patient refusal, infection at the puncture site and hemodynamic instability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of effectiveness of epidural morphine/ropivacaine treatment | Up to 60 days
  Change From Baseline in Pain Scores on the Visual Analog Scale (0 means no pain and 10 means worst pain) in patients in the control group and intervention group for up to 60 days.

SECONDARY OUTCOMES:
Assessment of quality of life | Up to 60 days
  Change of quality of life score by the European Organization for Research and Treatment of Cancer QLQ-C30 (EORTC QLQ-C30), which consists of a likert-type scale ranging from 1 to 4 for functions and symptoms, where 1= not at all, 2=slightly, 3= moderately, and 4 = very much. If the resulting score on the functional scale is high, this represents a healthy functional level, while a high score on the symptom scale represents a low level of symptom tolerance and treatment side effects. This scale also assesses overall health, ranging from 1 to 7, with 1=bad and 7 = very good
Assessment of functional status | Up to 60 days
  Change in the patient's functional status by the Karnofsky Performance Scale (KPS), which ranges from 100% to 0%, where 100% means no evidence of disease and 0% means death
Assessment of progression of disease status | Up to 60 days
  Change in disease status using the Eastern Cooperative Oncology Group (ECOG) scale, ranging from 0 to 5, where 0 = completely active and 5 =dead
Assessment of patient's clinical-functional status | Up to 60 days
  Change in clinical-functional status by the Palliative Performance Scale (PPS), which ranges from 100 to 0%, where 100% = good clinical-functional status and 0%= dead
Assessment of disease prognosis | Up to 60 days
  Change in survival time by the Palliative Prognosis Scale (PPI), which assesses PPS, presence of delirium, dyspnea, oral intake and edema, where each factor presents a score and at the end the scores are summed and the patient is classified into group A (Total Score < 2.0): > 6 weeks survival, group B (Total Score between 2.0 - 4.0): 3 - 6 weeks survival and group C (Total Score > 4.0): < 3 weeks survival
Cost-effectiveness analysis | Up to 60 days
  For cost-effectiveness analysis, a direct cost analysis using the cost-effectiveness ratio will be used. The costs considered in this study will be the direct non-medical and direct medical costs. For direct cost analysis, the microcosting technique will be used.
  For economic analysis, the incremental cost-effectiveness ratio (ICER) will be used. Once a CERI is obtained, the result is evaluated by defining a cost-effectiveness threshold, which aims to identify values that society considers feasible, from an economic point of view, to be incorporated as additional costs in society's spending on health (BRASIL, 2014).
  Once the RCEI is obtained, the next step in a pharmacoeconomic analysis will be to perform a sensitivity analysis of the parameters involved during the research.
Quantify the plasma concentration of morphine | Up to 60 days
  Patients will undergo blood draws to obtain plasma, 1:30h after taking morphine (oral or epidural) which will later be quantified for morphine by gas chromatography.
Correlating plasma morphine concentration with therapeutic effecs | Up to 60 days
  The amount of morphine found in plasma (outcome 8) will be correlated with the therapeutic effects (pain levels by Visual Analog Scale)
Quantify brain-derived neurotrophic factor (BDNF) | Up to 60 days
  BDNF quantification will be done in the plasma of the patients, using the BDNF enzyme-linked immunosorbent assay (ELISA) kit from sigma and adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Larissa LT Pacheco, PhD, Study Director — Universidade Federal de Alfenas
Locations (1):
- Larissa Helena Lobo Torres Pacheco, Alfenas, Minas Gerais, Brazil